CLINICAL TRIAL: NCT02500706
Title: Efficacy and Safety of Faster-acting Insulin Aspart Compared to NovoRapid® Both in Combination With Insulin Degludec in Adults With Type 1 Diabetes
Acronym: onset®8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-4131; 2015-001047-36 (EudraCT Number); U1111-1167-9495 (Other: WHO)
Record Dates: First submitted 2015-07-15; First posted 2015-07-16 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mealtime faster-acting insulin aspart and insulin degludec (Experimental)
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin degludec
- Mealtime NovoRapid® and insulin degludec (Active Comparator)
  Interventions: Drug: insulin aspart; Drug: insulin degludec
- Postmeal faster-acting insulin aspart and insulin degludec (Experimental)
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin degludec

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Injected subcutaneously (under the skin) three times daily for 26 weeks. Dose individually adjusted. Mealtime dosing is defined as injecting 0-2 minutes before the meal. Postmeal dosing is defined as injecting 20 minutes after the start of the meal.
  Arms: Mealtime faster-acting insulin aspart and insulin degludec; Postmeal faster-acting insulin aspart and insulin degludec
Drug: insulin aspart — Injected subcutaneously (under the skin) three times daily for 26 weeks. Dose individually adjusted. Mealtime dosing is defined as injecting 0-2 minutes before the meal.
  Arms: Mealtime NovoRapid® and insulin degludec
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily for 26 weeks. Dose individually adjusted

SUMMARY:
This trial is conducted in Asia, Europe and North America. The purpose is to confirm efficacy in terms of glycaemic control of treatment with mealtime faster-acting insulin aspart in combination with insulin degludec in adults with Type 1 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria: - Male or female, age greater than or equal to 18 years ( for Japan and Taiwan: age greater than or equal to 20 years) at the time of signing informed consent - Type 1 Diabetes Mellitus (based on clinical judgement and/or supported by laboratory analysis as per local guidelines) 12 months or more prior to screening - Currently treated with a basal-bolus insulin regimen for at least 12 months prior to screening (Visit 1) - Currently treated with a basal insulin analogue for at least 4 months prior to screening (Visit 1) - HbA1c 7.0-9.5% (53-80 mmol/mol) (both inclusive) as assessed by central laboratory - Body Mass Index less than or equal to 35.0 kg/m^2 Exclusion Criteria: - Within the past 180 days any of the following: myocardial infarction, stroke or hospitalization for unstable angina and/or transient ischemic attack - Subjects presently classified as being in New York Heart Association (NYHA) Class IV Currently planned coronary, carotid or peripheral artery revascularisation - Diabetic ketoacidosis requiring hospitalisation within the last 180 days prior to screening (Visit 1) - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of three months before screening (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (129):
- United States (52):
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, Newport Beach, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Hamilton, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Bend, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Beaumont, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Federal Way, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Bulgaria (6):
  - Novo Nordisk Investigational Site, Dimitrovgrad
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Canada (5):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Québec
- Germany (7):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Lingen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Schweinfurt
- India (14):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Rohtak, Haryana
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Chandigarh
  - Novo Nordisk Investigational Site, New Dehli
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Pune
- Israel (5):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
- Italy (6):
  - Novo Nordisk Investigational Site, Ancona
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Sesto San Giovanni (MI)
- Japan (20):
  - Novo Nordisk Investigational Site, Amagasaki-shi, Hyogo
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi, Kanagawa
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kobe-shi, Hyogo
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Matsumoto-shi, Nagano
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Russia (7):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Tyumen
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Taiwan (2):
  - Novo Nordisk Investigational Site, Taipei
  - Novo Nordisk Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Background] Rose L, Kadowaki T, Pieber TR, Buchholtz K, Ekelund M, Gorst-Rasmussen A, Philis-Tsimikas A. Efficacy and Safety of Fast-Acting Insulin Aspart in People with Type 1 Diabetes Using Carbohydrate Counting: A Post Hoc Analysis of Two Randomised Controlled Trials. Diabetes Ther. 2019 Jun;10(3):1029-1041. doi: 10.1007/s13300-019-0608-4. Epub 2019 Apr 4. PMID 30949906
- [Result] Buse JB, Carlson AL, Komatsu M, Mosenzon O, Rose L, Liang B, Buchholtz K, Horio H, Kadowaki T. Fast-acting insulin aspart versus insulin aspart in the setting of insulin degludec-treated type 1 diabetes: Efficacy and safety from a randomized double-blind trial. Diabetes Obes Metab. 2018 Dec;20(12):2885-2893. doi: 10.1111/dom.13545. Epub 2018 Oct 10. PMID 30259644
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 146 sites in 12 countries(number of sites indicates those that both screened and randomised subjects, unless otherwise noted)-Austria(4);Bulgaria(8); Canada(6); Germany(7); India(16); Israel(6); Italy(4); Japan(24); Russian Federation(10); Serbia(3); Taiwan(3); United States(55 sites screened/52 sites randomised subjects)
Pre-assignment Details: Eligible subjects were enrolled in a 8-week run-in period (1108 subjects) where subjects were switched from previous insulin treatment to insulin degludec once daily,and NovoRapid®/NovoLog® as mealtime bolus insulin. The basal insulin treatment was optimised using treat-to-target approach. 83 subjects were run-in failures and 1025 were randomised.
Groups:
- Faster Aspart (Meal): Bolus insulin: Participants received subcutaneous (s.c., into the abdominal wall) injections of faster-acting insulin aspart at mealtime (0-2 minutes before the meal) during 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the glycaemic target of pre-prandial and bedtime plasma glucose between 4.0-6.0 mmol/L (71-108 mg/dL) in a treat-to-target fashion.
  Basal insulin: Participants continued insulin degludec once daily s.c. injections at the dose optimized during run-in period during 26-week treatment period.
- Faster Aspart (Post): Bolus insulin: Participants received s.c. injections of faster-acting insulin aspart at mealtime (injecting the bolus insulin at the end of the meal but no later than 20 minutes after the start of the meal) during 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the glycaemic target of pre-prandial and bedtime plasma glucose between 4.0-6.0 mmol/L (71-108 mg/dL) in a treat-to-target fashion.
  Basal insulin: Participants continued insulin degludec once daily s.c. injections at the dose optimized during run-in period during 26-week treatment period.
- NovoRapid (Meal): After 8-week run-in period, subjects continued using mealtime insulin aspart (NovoRapid®/NovoLog®) s.c. injections at mealtime (0-2 minutes before the meal) during 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the glycaemic target of pre-prandial and bedtime plasma glucose between 4.0-6.0 mmol/L (71-108 mg/dL) in a treat-to-target fashion.
  Basal insulin: Participants continued insulin degludec once daily s.c. injections at the dose optimized during run-in period during 26-week treatment period.
Period: Overall Study
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Started | 342 | 341 | 342
Exposed | 342 | 341 | 342
Completed | 338 | 334 | 335
Not Completed | 4 | 7 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 6 | 4
Not completed — Unclassified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal) | Total
Number analyzed (Participants) | 342 | 341 | 342 | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.48 (14.42) | 41.02 (14.59) | 40.77 (14.22) | 41.09 (14.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 155 | 163 | 476
  Male | 184 | 186 | 179 | 549
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 12 | 33
  Not Hispanic or Latino | 329 | 333 | 330 | 992
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 116 | 131 | 137 | 384
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 6 | 16
  White | 219 | 206 | 198 | 623
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.46 (0.68) | 7.40 (0.60) | 7.41 (0.79) | 7.42 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c 26 Weeks After Randomisation
Description: Change from baseline (week 0) in HbA1c was evaluated after 26 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In-trial period: the observation period from date of randomisation until last trial-related subject-site contact.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of subjects analysed=subject with data available for HbA1c.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 341
percentage of HbA1c | -0.12 (0.64) | 0.005 (0.64) | -0.09 (0.65)
Statistical Analysis 1: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); The endpoint was analysed using an analysis of variance model after multiple imputation assuming treatment according to randomisation. The model includes treatment, region and bolus adjusting method at randomisation as factors, and baseline HbA1c as a covariate; Test type: Non-Inferiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 1: Primary analysis: HbA1c non-inferiority of mealtime faster aspart versus mealtime NovoRapid®/NovoLog®. Non-inferiority of mealtime faster aspart was considered confirmed if the upper boundary of the two-sided 95% CI was below or equal to 0.4%; p < 0.001, ANOVA model after multiple imputation — p-value from the 2-sided test for treatment difference evaluated at the 5% level; Treatment difference = -0.02, 95% CI 2-sided [-0.11 to 0.07]
Statistical Analysis 2: Comparison: Faster Aspart (Post) vs NovoRapid (Meal); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 2: HbA1c non-inferiority of postmeal faster aspart versus mealtime NovoRapid®/NovoLog®. Non-inferiority of postmeal faster aspart was considered confirmed if the upper boundary of the two-sided 95% CI was below or equal to 0.4%; p < 0.001, ANOVA model after multiple imputation — p-value from the 2-sided test for treatment difference evaluated at the 5% level; Treatment difference = 0.10, 95% CI 2-sided [0.004 to 0.19]
Statistical Analysis 3: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 4: HbA1c superiority of mealtime faster aspart versus mealtime NovoRapid®/NovoLog®. Superiority was to be confirmed if the upper boundary of the two-sided 95% CI of the mean treatment difference (mealtime faster aspart minus mealtime NovoRapid®/NovoLog®) was below 0%-points; p = 0.633, ANOVA model after multiple imputation — p-value from the 2-sided test for treatment difference evaluated at the 5% level; Treatment difference = -0.02, 95% CI 2-sided [-0.11 to 0.07]

2. Secondary Outcome: Change From Baseline in 1-hour Post Prandial Glucose (PPG) Increment 26 Weeks After Randomisation (Meal Test)
Description: The 1-hour PPG increment was analysed based on the laboratory-measured values in the meal test, and was derived using the 1-hour PPG measurement minus the pre-prandial plasma glucose (PG). The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of subjects analysed=subject with data available for 1-hour PPG and pre-prandial PG.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 332 | 332 | 326
mmol/L | -1.13 (4.04) | 1.04 (3.53) | -0.15 (3.78)
Statistical Analysis 1: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); Change from baseline in postprandial glucose increment (meal test) is analysed using an analysis of variance model. The model includes treatment, region and bolus adjusting method at randomisation as factors, and baseline postprandial glucose increment as a covariate; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 3: 1-hour postprandial glucose (PPG) increments superiority of mealtime faster aspart versus mealtime NovoRapid®/NovoLog. Superiority was confirmed if the upper boundary of the two-sided 95% CI of the mean treatment difference (mealtime faster aspart minus mealtime NovoRapid®/NovoLog®) was below 0; p < 0.001, ANOVA — p-value from the 2-sided test for treatment difference evaluated at the 5% level; Treatment difference = -0.90, 95% CI 2-sided [-1.36 to -0.45]

3. Secondary Outcome: Change From Baseline in 1,5-anhydroglucitol 26 Weeks After Randomisation
Description: The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of subjects analysed=subject with data available for 1,5-anhydroglucitol.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 341 | 336 | 338
ug/mL | 0.22 (2.23) | -0.15 (2.10) | 0.22 (2.25)
Statistical Analysis 1: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); Change from baseline in 1,5-anhydroglucitol was analysed using an analysis of variance model after multiple imputation assuming treatment according to randomisation. The model includes treatment, region and bolus adjusting method at randomisation as factors, and baseline 1,5-anhydroglucitol as a covariate; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 5: 1,5-anhydroglucitol superiority of mealtime faster aspart versus mealtime NovoRapid®/NovoLog®. Superiority was to be confirmed if the lower boundary of the two-sided 95% CI of the mean treatment difference (mealtime faster aspart minus mealtime NovoRapid®/NovoLog®) was above 0; p = 0.924, ANOVA model after multiple imputation — p-values are from the 2-sided test for treatment difference evaluated at the 5% level; Treatment difference = 0.02, 95% CI 2-sided [-0.31 to 0.34]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) 26 Weeks After Randomisation
Description: The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of subjects analysed=subject with data available for HbA1c.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 339 | 338 | 336
mmol/L | 0.17 (2.94) | 0.44 (3.29) | 0.64 (3.35)

5. Secondary Outcome: Percentage of Subjects Reaching HbA1c Targets (HbA1c < 7.0%) 26 Weeks After Randomisation
Description: The percentage of subjects who achieved the HbA1c target of <7.0% 26 weeks after randomisation. Subjects without an HbA1c measurement at week 26 were treated as non-responders.
Time Frame: 26 weeks after randomisation
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Yes | 28.7 | 28.2 | 32.7
  No | 71.3 | 71.8 | 67.3

6. Secondary Outcome: Percentage of Subjects Reaching HbA1c Targets (HbA1c < 7.0% Without Severe Hypoglycaemia) 26 Weeks After Randomisation
Description: The percentage of subjects who achieved the HbA1c target of <7.0% without severe hypoglycaemia 26 weeks after randomisation. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Subjects without an HbA1c measurement at week 26 were treated as non-responders.
Time Frame: 26 weeks after randomisation
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Yes | 25.7 | 26.4 | 30.4
  No | 74.3 | 73.6 | 69.6

7. Secondary Outcome: Percentage of Subjects Reaching HbA1c Targets (HbA1c < 7.0% Without Severe Hypoglycaemia and Minimal Weight Gain [<3.0%]) 26 Weeks After Randomisation
Description: The percentage of subjects who achieved the HbA1c target of <7.0% without severe hypoglycaemia and with minimal weight gain (defined as less than a 3% increase) 26 weeks after randomisation. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Subjects without an HbA1c measurement at week 26 or without body weight measurement at week 26 were treated as non-responders.
Time Frame: 26 weeks after randomisation
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Yes | 16.4 | 17.9 | 19.3
  No | 83.6 | 82.1 | 80.7

8. Secondary Outcome: Change From Baseline in 30- Min, 1- Hour, 2- Hour, 3- Hour and 4- Hour PPG 26 Weeks After Randomisation
Description: Laboratory measured PG from the meal test was analysed for 30, 60, 120, 180, and 240 minutes PPG separately. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subject with data available for PPG at individual timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
mmol/L
  Change in PPG at 30 min: number analyzed (Participants) | 333 | 331 | 326
  Change in PPG at 30 min | -0.47 (3.58) | 1.31 (3.52) | 0.21 (3.78)
  Change in PPG at 1 hour: number analyzed (Participants) | 333 | 333 | 326
  Change in PPG at 1 hour | -1.05 (4.56) | 1.39 (4.44) | 0.20 (4.52)
  Change in PPG at 2 hours: number analyzed (Participants) | 329 | 333 | 323
  Change in PPG at 2 hours | -0.41 (5.17) | 0.80 (5.38) | 0.33 (5.51)
  Change in PPG at 3 hours: number analyzed (Participants) | 332 | 327 | 324
  Change in PPG at 3 hours | -0.12 (5.20) | 0.93 (5.06) | 0.51 (5.33)
  Change in PPG at 4 hours: number analyzed (Participants) | 330 | 328 | 325
  Change in PPG at 4 hours | 0.005 (4.64) | 0.83 (4.59) | 0.53 (4.60)

9. Secondary Outcome: Change From Baseline in 30- Min, 1- Hour, 2- Hour, 3- Hour and 4- Hour PPG Increment 26 Weeks After Randomisation
Description: Laboratory measured PG from the meal test was analysed for 30, 60, 120, 180, and 240 minutes PPG separately. The corresponding PPG increments were derived separately using each PPG measurement minus the pre-prandial PG. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subject with data available for PPG and pre-prandial PG at individual timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
mmol/L
  Change in PPG increment at 30 min: number analyzed (Participants) | 332 | 330 | 326
  Change in PPG increment at 30 min | -0.55 (2.55) | 0.94 (2.47) | -0.14 (2.63)
  Change in PPG increment at 1 hour: number analyzed (Participants) | 332 | 332 | 326
  Change in PPG increment at 1 hour | -1.13 (4.04) | 1.04 (3.53) | -0.15 (3.78)
  Change in PPG increment at 2 hours: number analyzed (Participants) | 328 | 331 | 323
  Change in PPG increment at 2 hours | -0.47 (4.74) | 0.42 (5.01) | -0.01 (5.15)
  Change in PPG increment at 3 hours: number analyzed (Participants) | 331 | 326 | 324
  Change in PPG increment at 3 hours | -0.20 (4.89) | 0.55 (4.95) | 0.11 (5.32)
  Change in PPG increment at 4 hours: number analyzed (Participants) | 329 | 327 | 325
  Change in PPG increment at 4 hours | -0.10 (4.47) | 0.45 (4.44) | 0.16 (4.63)

10. Secondary Outcome: Change From Baseline in 7-9-7-point Self-measured Plasma Glucose (SMPG) 26 Weeks After Randomisation: Mean of the 7-9-7-point Profile
Description: The subject was instructed to perform a 7-9-7 SMPG point profile on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. The mean of the 7-9-7-point profile was defined as the area under the curve profile divided by the measurement time, and was calculated using the linear trapezoidal technique. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subject with data available for 7-9-7 point profile.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 320 | 327 | 320
mmol/L | -0.304 (1.928) | -0.231 (1.846) | -0.309 (2.060)

11. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG 26 Weeks After Randomisation: PPG (Mean, Breakfast, Lunch, Main Evening Meal)
Description: The subject was instructed to perform a 7-9-7 SMPG point profile on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. Results were derived from the three profiles: post-breakfast, post-lunch, post-main evening meal. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subject with data available data at three profiles: post-breakfast, post-lunch, post-main evening meal.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
mmol/L
  Change in PPG breakfast: number analyzed (Participants) | 313 | 326 | 316
  Change in PPG breakfast | -0.83 (3.34) | -0.03 (3.30) | -0.31 (3.18)
  Change in PPG lunch: number analyzed (Participants) | 313 | 323 | 318
  Change in PPG lunch | -0.59 (3.04) | 0.06 (2.98) | -0.33 (3.38)
  Change in PPG main evening meal: number analyzed (Participants) | 314 | 321 | 319
  Change in PPG main evening meal | -0.53 (3.55) | -0.01 (3.56) | -0.14 (3.22)
  Change in PPG all meals: number analyzed (Participants) | 308 | 317 | 313
  Change in PPG all meals | -0.65 (2.26) | -0.004 (2.19) | -0.25 (2.33)

12. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG 26 Weeks After Randomisation: PPG Increment (Mean, Breakfast, Lunch, Main Evening Meal)
Description: The subject was instructed to perform a 7-9-7 SMPG point profile on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. PPG increment for each meal (breakfast, lunch, main evening meal) was derived from the 7-point and 9-point profile as the difference between PPG values and the PG value before the meal in each separate profile. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subject with data available data for PPG values and the PG value before the meal (breakfast, lunch, main evening meal).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
mmol/L
  Change in PPG increment breakfast: number analyzed (Participants) | 313 | 326 | 316
  Change in PPG increment breakfast | -1.14 (3.64) | 0.06 (3.51) | -0.30 (3.16)
  Change in PPG increment lunch: number analyzed (Participants) | 313 | 321 | 317
  Change in PPG increment lunch | -0.67 (3.20) | -0.08 (3.10) | -0.004 (3.31)
  Change in PPG increment main evening meal: number analyzed (Participants) | 313 | 320 | 319
  Change in PPG increment main evening meal | -0.29 (3.70) | 0.34 (3.54) | 0.26 (3.49)
  Change in PPG increment all meals: number analyzed (Participants) | 307 | 315 | 313
  Change in PPG increment all meals | -0.72 (2.06) | 0.08 (1.98) | -0.02 (2.01)

13. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG 26 Weeks After Randomisation: Fluctuation in 7-9-7-point Profile
Description: The subject was instructed to perform a 7-9-7 SMPG point profile on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. Fluctuation in SMPG profile was the average absolute difference from the mean of the SMPG profile. Change from baseline is represented as ratio to baseline value. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subjects who contributed to this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 331 | 335 | 331
ratio | 0.876 (47.490) | 0.875 (40.293) | 0.890 (41.978)

14. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG 26 Weeks After Randomisation: Change in the Nocturnal Self-measured Plasma Glucose Measurements
Description: The subject was instructed to perform 7-9-7 SMPG point profile on 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast,60 minutes after the start of breakfast,before lunch,60 minutes after the start of lunch, before main evening meal,60 minutes after the start of main evening meal,and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on following day. Change from baseline in nocturnal PG values (nocturnal increments) was assessed by considering differences between PG values available at bedtime, at 4 a.m and the before breakfast value the following day: (04:00 PG value minus at bedtime PG value), (before breakfast PG value minus at bedtime PG value) and (before breakfast PG value minus 04:00 PG value). Results are based on the last in-trial value (the last available measurement in the in-trial period).
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number of analysed=subjects with available data for nocturnal SMPG measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
mmol/L
  Change in nocturnal increment-bedtime to 04:00: number analyzed (Participants) | 178 | 208 | 188
  Change in nocturnal increment-bedtime to 04:00 | 0.14 (5.66) | 0.19 (6.41) | 0.45 (5.55)
  Change in nocturnal increment-bedtime to breakfast: number analyzed (Participants) | 274 | 278 | 278
  Change in nocturnal increment-bedtime to breakfast | 0.86 (6.21) | 0.93 (6.24) | 0.33 (5.71)
  Change in nocturnal increment-04:00 to breakfast: number analyzed (Participants) | 176 | 209 | 191
  Change in nocturnal increment-04:00 to breakfast | 0.78 (4.95) | 1.01 (4.12) | -0.02 (4.17)

15. Secondary Outcome: Percentage of Subjects Reaching PPG Target (Overall Mean of Daily PPG Measurements in SMPG) 26 Weeks After Randomisation: Overall PPG (1 Hour) ≤7.8 mmol/L
Description: Percentage of subjects achieving an overall mean 1-hour PPG ≤7.8 mmol/L [140 mg/dL] 26 weeks after randomisation. Subjects without an overall mean 1-hour PPG at week 26 were treated as non-responders.
Time Frame: 26 weeks after randomisation
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Yes | 27.8 | 19.9 | 21.6
  No | 72.2 | 80.1 | 78.4

16. Secondary Outcome: Percentage of Subjects Reaching PPG Target (Overall Mean of Daily PPG Measurements in SMPG) 26 Weeks After Randomisation: Overall PPG (1 Hour) ≤7.8 mmol/L Without Severe Hypoglycaemia
Description: Percentage of subjects achieving an overall mean 1-hour PPG ≤7.8 mmol/L [140 mg/dL] 26 weeks after randomisation without severe hypoglycaemia. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Subjects without an overall mean 1-hour PPG at week 26 were treated as non-responders.
Time Frame: 26 weeks after randomisation
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Yes | 24.6 | 18.8 | 20.5
  No | 75.4 | 81.2 | 79.5

17. Secondary Outcome: Percentage of Subjects Reaching PPG Target (Overall Mean of Daily PPG Measurements in SMPG) 26 Weeks After Randomisation: Overall PPG (1 Hour) ≤7.8 mmol/L and HbA1c <7.0% and Minimal Weight Gain (<3.0%) Without Severe Hypoglycaemia
Description: The percentage of subjects who achieved overall mean 1 hour PPG ≤7.8 mmol/L [140 mg/dL], had HbA1c < 7.0% and had minimal weight gain (increase in body weight from baseline <3.0%) 26 weeks after randomisation, and without severe hypoglycaemic episodes. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Subjects without an overall mean 1-hour PPG or an HbA1c value or a body weight at week 26 were treated as non-responders.
Time Frame: 26 weeks after randomisation
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Yes | 7.6 | 4.7 | 8.2
  No | 92.4 | 95.3 | 91.8

18. Secondary Outcome: Change From Baseline in Lipids-lipoproteins Profile 26 Weeks After Randomisation (Total Cholesterol, High Density Lipoproteins [HDL] Cholesterol, Low Density Lipoproteins [LDL] Cholesterol)
Description: Change from baseline in HDL cholesterol, LDL cholesterol and total cholesterol 26 weeks after randomization are represented as ratio to baseline values. The results are based on the last in-trial value (the last available measurement in the in-trial period).
Time Frame: Week 0, week 26
Population: Analysis was based on FAS. Number analysed=number of subjects with available data for individual lipid parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
ratio
  HDL cholesterol: number analyzed (Participants) | 340 | 340 | 341
  HDL cholesterol | 0.981 (16.200) | 0.998 (17.283) | 0.999 (33.056)
  LDL cholesterol: number analyzed (Participants) | 340 | 340 | 341
  LDL cholesterol | 1.025 (20.067) | 1.053 (22.465) | 1.062 (215.570)
  Total cholesterol: number analyzed (Participants) | 340 | 340 | 341
  Total cholesterol | 1.002 (14.561) | 1.030 (15.789) | 1.020 (15.891)

19. Secondary Outcome: Insulin Dose (Basal Insulin Dose, Total and Individual Meal Insulin Dose)
Description: The insulin doses were summarised descriptively at week 0 and week 26 both by meal type and as total daily dose (total daily and separately for each mealtime dose). Week 26 results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on safety analysis set (all subjects receiving at least one dose of the investigational product or its comparator). Number of subjects analysed=subjects with available data for specified categories.
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
Units
  Daily bolus insulin dose: week 0: number analyzed (Participants) | 339 | 336 | 335
  Daily bolus insulin dose: week 0 | 25.5 (15.4) | 25.4 (14.3) | 26.6 (14.8)
  Daily bolus insulin dose: Last on-treatment value: number analyzed (Participants) | 341 | 337 | 340
  Daily bolus insulin dose: Last on-treatment value | 31.1 (19.4) | 30.5 (18.9) | 33.5 (22.5)
  Daily basal insulin dose: week 0: number analyzed (Participants) | 342 | 339 | 339
  Daily basal insulin dose: week 0 | 25.3 (14.5) | 26.7 (15.6) | 26.2 (15.0)
  Daily basal insulin dose: Last on-treatment value: number analyzed (Participants) | 342 | 339 | 340
  Daily basal insulin dose: Last on-treatment value | 26.7 (16.6) | 27.3 (16.8) | 27.2 (17.3)
  Total daily insulin dose: week 0: number analyzed (Participants) | 339 | 335 | 335
  Total daily insulin dose: week 0 | 50.8 (26.1) | 52.2 (25.2) | 53.1 (25.9)
  Total daily insulin dose: Last on-treatment value: number analyzed (Participants) | 341 | 336 | 340
  Total daily insulin dose: Last on-treatment value | 57.7 (31.4) | 57.8 (30.2) | 60.4 (34.0)
  Daily breakfast bolus insulin dose: Last value: number analyzed (Participants) | 341 | 340 | 340
  Daily breakfast bolus insulin dose: Last value | 8.8 (6.2) | 8.6 (6.0) | 9.5 (7.7)
  Daily lunch bolus insulin dose: Last value: number analyzed (Participants) | 342 | 340 | 340
  Daily lunch bolus insulin dose: Last value | 10.5 (7.0) | 10.3 (6.9) | 11.2 (7.6)
  Daily main evening meal bolus insulin: Last value: number analyzed (Participants) | 342 | 340 | 340
  Daily main evening meal bolus insulin: Last value | 11.9 (7.7) | 11.6 (7.4) | 12.7 (9.1)
  Daily other bolus insulin dose: Last value: number analyzed (Participants) | 166 | 167 | 153
  Daily other bolus insulin dose: Last value | 4.7 (5.1) | 4.3 (3.5) | 4.2 (3.3)

20. Secondary Outcome: Number of Treatment Emergent Adverse Events During 26 Weeks After Randomisation
Description: A treatment emergent adverse event (TEAE) was defined as an event that had an onset date on or after the first day of exposure to randomised treatment, and no later than seven days after the last day of randomised treatment.
Time Frame: Week 0 to week 26 (+7 days)
Population: Analysis was based on SAS.
Measure: Number; unit: events
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
events | 649 | 656 | 627

21. Secondary Outcome: Number of Treatment-emergent Injection Site Reactions During the 26 Weeks After Randomisation
Description: A treatment emergent event was defined as an event that had an onset date on or after the first day of exposure to randomised treatment, and no later than seven days after the last day of randomised treatment.
Time Frame: Week 0 to week 26 (+7 days)
Population: Analysis was based on SAS.
Measure: Number; unit: Injection site reactions
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
Injection site reactions | 9 | 12 | 10

22. Secondary Outcome: Number of Hypoglycaemic Episodes Classified Both According to the American Diabetes Association (ADA) Definition and Novo Nordisk (NN) Definition During 26 Weeks After Randomisation: Overall
Description: ADA classification includes following criteria: Severe,Documented symptomatic,Asymptomatic,Probable symptomatic,Pseudo-hypoglycaemia.
  NN Classification:
  * Severe:same as per ADA classification
  * Symptomatic blood glucose (BG) confirmed: PG<3.1 mmol/L with symptoms consistent with hypoglycaemia
  * Asymptomatic BG confirmed:PG<3.1 mmol/L without symptoms consistent with hypoglycaemia
  * Severe or BG confirmed symptomatic:severe according to ADA classification or BG confirmed by PG<3.1 mmol/L with symptoms consistent with hypoglycaemia
  * BG confirmed:PG<3.1 mmol/L with or without symptoms consistent with hypoglycaemia
  * Severe or BG confirmed:severe according to ADA classification or BG confirmed by PG<3.1 mmol/L with or without symptoms consistent with hypoglycaemia
  * Unclassifiable Results represent total number of hypoglycaemic episodes. Treatment emergent episode: an event that has onset up to 1 day after last day of randomised treatment and excluding events occurring in run-in period.
Time Frame: Week 0 to week 26 (+1 day)
Population: Analysis was based on SAS.
Measure: Number; unit: hypoglycaemic episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
hypoglycaemic episodes | 15760 | 16579 | 16520

23. Secondary Outcome: Number of Hypoglycaemic Episodes Classified Both According to the ADA Definition and Novo Nordisk Definition During 26 Weeks After Randomisation: Daytime and Nocturnal Hypoglycaemic Episodes (00:01-05:59 - Inclusive)
Description: ADA classification includes following criteria: Severe, Documented symptomatic, Asymptomatic, Probable symptomatic, Pseudo-hypoglycaemia.
  NN Classification:
  * Severe: same as per ADA classification
  * Symptomatic BG confirmed: PG<3.1 mmol/L with symptoms consistent with hypoglycaemia
  * Asymptomatic BG confirmed: PG<3.1 mmol/L without symptoms consistent with hypoglycaemia
  * Severe or BG confirmed symptomatic: severe according to the ADA classification or BG confirmed by PG<3.1 mmol/Lwith symptoms consistent with hypoglycaemia
  * BG confirmed: PG<3.1 mmol/L with or without symptoms consistent with hypoglycaemia
  * Severe or BG confirmed: severe according to the ADA classification or BG confirmed by PG<3.1 mmol/L with or without symptoms consistent with hypoglycaemia
  * Unclassifiable Results represent total number of hypoglycaemic episodes. Nocturnal hypoglycaemic episodes were episodes occurring between 00:01 and 05:59 both inclusive.
Time Frame: Week 0 to week 26 (+1 day)
Population: Analysis was based on SAS.
Measure: Number; unit: hypoglycaemic episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
hypoglycaemic episodes
  Daytime hypoglycaemic episodes | 14570 | 15379 | 15257
  Nocturnal hypoglycaemic episodes | 1190 | 1200 | 1263

24. Secondary Outcome: Number of Hypoglycaemic Episodes Classified Both According to the ADA Definition and Novo Nordisk Definition During 26 Weeks After Randomisation: From Start of Meal Until 1,2, 4 Hours and From 2 Hours (Exclusive) to 4 Hours (Inclusive) After Start of Meal
Description: ADA classification includes following criteria: Severe, Documented symptomatic, Asymptomatic, Probable symptomatic, Pseudo-hypoglycaemia.
  NN Classification:
  * Severe: same as per ADA classification
  * Symptomatic BG confirmed: PG<3.1 mmol/L with symptoms consistent with hypoglycaemia
  * Asymptomatic BG confirmed: PG<3.1 mmol/L without symptoms consistent with hypoglycaemia
  * Severe or BG confirmed symptomatic: severe according to the ADA classification or BG confirmed by PG<3.1 mmol/Lwith symptoms consistent with hypoglycaemia
  * BG confirmed: PG<3.1 mmol/L with or without symptoms consistent with hypoglycaemia
  * Severe or BG confirmed: severe according to the ADA classification or BG confirmed by PG<3.1 mmol/L with or without symptoms consistent with hypoglycaemia
  * Unclassifiable Results represent total number of hypoglycaemic episodes related to meals.
Time Frame: Week 0 to week 26 (+1 day)
Population: Analysis was based on SAS.
Measure: Number; unit: hypoglycaemic episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
hypoglycaemic episodes
  Within 1 hour after meal | 624 | 614 | 459
  Within 2 hours after meal | 1314 | 1470 | 1224
  Within 4 hours after meal | 3920 | 4794 | 4129
  Between 1 (exclusive) to 2 hours (inclusive) | 690 | 856 | 765
  Between 2 (exclusive) to 3 hours (inclusive) | 1236 | 1634 | 1302
  Between 2 (exclusive) to 4 hours (inclusive) | 2606 | 3324 | 2905
  Between 3 (exclusive) to 4 hours (inclusive) hours | 1370 | 1690 | 1603

25. Secondary Outcome: Change From Baseline 26 Weeks After Randomisation in Clinical Evaluations (Physical Examination)
Description: The physical examination parameters included head, ears, eyes, nose, throat, neck; respiratory system; cardiovascular system; gastrointestinal system including mouth; musculoskeletal system; central and peripheral nervous system; and skin. The examinations were measured as 'normal', 'abnormal, not clinically significant' (Abn, NCS) or 'abnormal, clinically significant' (Abn, CS). Reported results are percentage of subjects with 'normal', 'Abn, NCS' and 'Abn, CS' physical examinations at week 0 and week 26. Week 26 results are based on the last on-treatment value (last value), which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number analysed=number of subjects with available data for physical examinations at specified timepoints.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Cardiovascular system - Week 0: Normal | 97.4 | 98.8 | 97.7
  Cardiovascular system - Week 0: Abn, NCS | 2.6 | 0.9 | 2.0
  Cardiovascular system - Week 0: Abn, CS | 0.0 | 0.3 | 0.3
  Cardiovascular system - Last value: Normal: number analyzed (Participants) | 340 | 340 | 340
  Cardiovascular system - Last value: Normal | 97.4 | 98.8 | 97.9
  Cardiovascular system - Last value: Abn, NCS: number analyzed (Participants) | 340 | 340 | 340
  Cardiovascular system - Last value: Abn, NCS | 2.6 | 0.9 | 1.8
  Cardiovascular system - Last value: Abn, CS: number analyzed (Participants) | 340 | 340 | 340
  Cardiovascular system - Last value: Abn, CS | 0.0 | 0.3 | 0.3
  Nervous system - Week 0: Normal | 83.9 | 86.8 | 86.3
  Nervous system - Week 0: Abn, NCS | 15.5 | 12.9 | 13.2
  Nervous system - Week 0: Abn, CS | 0.6 | 0.3 | 0.6
  Nervous system - Last value: Normal: number analyzed (Participants) | 340 | 340 | 340
  Nervous system - Last value: Normal | 83.8 | 87.1 | 86.8
  Nervous system - Last value: Abn, NCS: number analyzed (Participants) | 340 | 340 | 340
  Nervous system - Last value: Abn, NCS | 15.6 | 12.9 | 12.4
  Nervous system - Last value: Abn, CS: number analyzed (Participants) | 340 | 340 | 340
  Nervous system - Last value: Abn, CS | 0.6 | 0.0 | 0.9
  Gastrointestinal system-week 0: Normal | 99.7 | 98.8 | 98.2
  Gastrointestinal system-week 0: Abn, NCS | 0.3 | 0.9 | 0.9
  Gastrointestinal system-week 0: Abn, CS | 0.0 | 0.3 | 0.9
  Gastrointestinal system-Last value: Normal: number analyzed (Participants) | 340 | 340 | 340
  Gastrointestinal system-Last value: Normal | 99.1 | 97.9 | 98.5
  Gastrointestinal system-Last value: Abn, NCS: number analyzed (Participants) | 340 | 340 | 340
  Gastrointestinal system-Last value: Abn, NCS | 0.9 | 1.2 | 0.6
  Gastrointestinal system-Last value: Abn, CS: number analyzed (Participants) | 340 | 340 | 340
  Gastrointestinal system-Last value: Abn, CS | 0.0 | 0.9 | 0.9
  Head,ears,eyes,nose,throat,neck:week 0-Normal | 95.0 | 95.6 | 93.3
  Head,ear,eye,nose,throat,neck-week 0:Abn,NCS | 4.1 | 3.8 | 5.8
  Head,ears,eyes,nose,throat,neck-week 0:Abn,CS | 0.9 | 0.6 | 0.9
  Head,ears,eyes,nose,throat,neck-Last value:Normal: number analyzed (Participants) | 340 | 340 | 340
  Head,ears,eyes,nose,throat,neck-Last value:Normal | 95.3 | 92.9 | 94.1
  Head,ear,eye,nose,throat,neck-Last value:Abn,NCS: number analyzed (Participants) | 340 | 340 | 340
  Head,ear,eye,nose,throat,neck-Last value:Abn,NCS | 3.8 | 6.2 | 4.4
  Head,ear,eye,nose,throat,neck-Last value:Abn,CS: number analyzed (Participants) | 340 | 340 | 340
  Head,ear,eye,nose,throat,neck-Last value:Abn,CS | 0.9 | 0.9 | 1.5
  Musculoskeletal system-week 0: Normal | 95.9 | 97.1 | 96.2
  Musculoskeletal system-week 0: Abn, NCS | 4.1 | 2.9 | 3.5
  Musculoskeletal system-week 0: Abn, CS | 0.0 | 0.0 | 0.3
  Musculoskeletal system-Last value: Normal: number analyzed (Participants) | 340 | 340 | 340
  Musculoskeletal system-Last value: Normal | 96.8 | 97.4 | 95.3
  Musculoskeletal system-Last value: Abn, NCS: number analyzed (Participants) | 340 | 340 | 340
  Musculoskeletal system-Last value: Abn, NCS | 3.2 | 2.6 | 3.8
  Musculoskeletal system-Last value: Abn, CS: number analyzed (Participants) | 340 | 340 | 340
  Musculoskeletal system-Last value: Abn, CS | 0.0 | 0.0 | 0.9
  Respiratory system-week 0: Normal | 99.4 | 99.4 | 99.1
  Respiratory system-week 0: Abn, NCS | 0.6 | 0.3 | 0.6
  Respiratory system-week 0: Abn, CS | 0.0 | 0.3 | 0.3
  Respiratory system-Last value: Normal: number analyzed (Participants) | 340 | 340 | 340
  Respiratory system-Last value: Normal | 99.7 | 99.4 | 99.4
  Respiratory system-Last value: Abn, NCS: number analyzed (Participants) | 340 | 340 | 340
  Respiratory system-Last value: Abn, NCS | 0.3 | 0.3 | 0.3
  Respiratory system-Last value: Abn, CS: number analyzed (Participants) | 340 | 340 | 340
  Respiratory system-Last value: Abn, CS | 0.0 | 0.3 | 0.3
  Skin-week 0: Normal | 91.5 | 89.7 | 91.5
  Skin-week 0: Abn, NCS | 7.3 | 8.8 | 7.9
  Skin-week 0: Abn, CS | 1.2 | 1.5 | 0.6
  Skin-Last value: Normal: number analyzed (Participants) | 340 | 340 | 340
  Skin-Last value: Normal | 91.5 | 91.5 | 92.4
  Skin-Last value: Abn, NCS: number analyzed (Participants) | 340 | 340 | 340
  Skin-Last value: Abn, NCS | 7.6 | 6.2 | 6.5
  Skin-Last value: Abn, CS: number analyzed (Participants) | 340 | 340 | 340
  Skin-Last value: Abn, CS | 0.9 | 2.4 | 1.2

26. Secondary Outcome: Change From Baseline in Blood Pressure 26 Weeks After Randomisation
Description: Change from baseline in systolic blood pressure and diastolic blood pressure 26 weeks after randomisation. Results are based on the last on-treatment value, which contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number of subjects analysed=subjects with available data for blood pressure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
mmHg
  Diastolic blood pressure | 0.5 (8.3) | 0.2 (7.8) | 0.8 (7.9)
  Systolic blood pressure | 0.6 (12.5) | 1.4 (10.8) | 0.8 (12.9)

27. Secondary Outcome: Change From Baseline in Pulse 26 Weeks After Randomisation
Description: Results are based on the last on-treatment value, which contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number of subjects analysed=subjects with available data for pulse.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
beats/minute | 0.0 (8.8) | -0.7 (9.3) | 0.7 (8.3)

28. Secondary Outcome: Change From Baseline in Clinical Evaluation (Electrocardiogram) 26 Weeks After Randomisation
Description: The electrocardiogram was interpreted by the investigator into following categories: Normal; Abn, NCS; Abnormal, CS. Reported results are percentage of subjects with 'normal', 'Abn, NCS' and 'Abn, CS' physical examinations at week 0 and week 26. Week 26 data are based on the last on-treatment value which contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number analysed=number of subjects with available data for electrocardiogram at specified timepoints.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Week 0: Normal | 80.7 | 81.8 | 84.2
  Week 0: Abn, NCS | 19.3 | 17.6 | 15.8
  Week 0: Abn, CS | 0.0 | 0.6 | 0.0
  Last on-treatment value: Normal: number analyzed (Participants) | 339 | 338 | 333
  Last on-treatment value: Normal | 80.8 | 84.0 | 82.3
  Last on-treatment value: Abn, NCS: number analyzed (Participants) | 339 | 338 | 333
  Last on-treatment value: Abn, NCS | 19.2 | 15.1 | 17.1
  Last on-treatment value: Abn, CS: number analyzed (Participants) | 339 | 338 | 333
  Last on-treatment value: Abn, CS | 0.0 | 0.9 | 0.6

29. Secondary Outcome: Change From Baseline in Clinical Evaluation (Fundoscopy/Fundus Photography) 26 Weeks After Randomisation
Description: The result of the fundus photography/dilated fundoscopy was interpreted by the investigator into following categories: Normal; Abn, NCS; Abnormal, CS. Reported results are percentage of subjects with 'normal', 'Abn, NCS' and 'Abn, CS' fundoscopy/fundus photography results at week 0 and week 26. Week 26 data are based on the last on-treatment value which contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number analysed=number of subjects with available data for fundoscopy/fundus photography at specified timepoints.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Left eye-Week 0: Normal | 65.8 | 68.0 | 69.3
  Left eye-Week 0: Abn, NCS | 26.9 | 23.5 | 23.4
  Left eye-Week 0: Abn, CS | 7.3 | 8.5 | 7.3
  Left eye-Last on-treatment value: Normal: number analyzed (Participants) | 333 | 333 | 332
  Left eye-Last on-treatment value: Normal | 62.5 | 69.4 | 69.3
  Left eye-Last on-treatment value: Abn, NCS: number analyzed (Participants) | 333 | 333 | 332
  Left eye-Last on-treatment value: Abn, NCS | 29.7 | 21.0 | 21.1
  Left eye-Last on-treatment value: Abn, CS: number analyzed (Participants) | 333 | 333 | 332
  Left eye-Last on-treatment value: Abn, CS | 7.8 | 9.6 | 9.6
  Right eye-Week 0: Normal | 65.2 | 68.9 | 67.0
  Right eye-Week 0: Abn, NCS | 27.8 | 22.3 | 25.4
  Right eye-Week 0: Abn, CS | 7.0 | 8.8 | 7.6
  Right eye-Last on-treatment value: Normal: number analyzed (Participants) | 333 | 333 | 332
  Right eye-Last on-treatment value: Normal | 64.0 | 67.9 | 68.7
  Right eye-Last on-treatment value: Abn, NCS: number analyzed (Participants) | 333 | 333 | 332
  Right eye-Last on-treatment value: Abn, NCS | 29.1 | 22.5 | 22.6
  Right eye-Last on-treatment value: Abn, CS: number analyzed (Participants) | 333 | 333 | 332
  Right eye-Last on-treatment value: Abn, CS | 6.9 | 9.6 | 8.7

30. Secondary Outcome: Change From Baseline in Erythrocytes 26 Weeks After Randomisation
Description: Week 26 data are based on the last on-treatment value, which contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for erythrocytes measurement.
Measure: Mean (Standard Deviation); unit: number of erythrocytes 10^12/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
number of erythrocytes 10^12/L | -0.01 (0.24) | -0.03 (0.26) | -0.02 (0.26)

31. Secondary Outcome: Change From Baseline in Haematocrit 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for haematocrit measurement.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
percentage of red blood cells in blood | -0.48 (2.58) | -0.52 (2.41) | -0.57 (2.45)

32. Secondary Outcome: Change From Baseline in Haemoglobin 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for haemoglobin measurement.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
mmol/L | -0.04 (0.51) | -0.04 (0.46) | -0.05 (0.50)

33. Secondary Outcome: Change From Baseline in Leukocytes 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for leukocytes measurement.
Measure: Mean (Standard Deviation); unit: Number of leukocytes 10^9/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
Number of leukocytes 10^9/L | -0.17 (1.63) | -0.03 (1.52) | -0.01 (1.46)

34. Secondary Outcome: Change From Baseline in Thrombocytes 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for thrombocytes measurement.
Measure: Mean (Standard Deviation); unit: Number of thrombocytes 10^9/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 339
Number of thrombocytes 10^9/L | -0.7 (40.0) | -2.0 (36.3) | -1.8 (33.7)

35. Secondary Outcome: Change From Baseline in Alanine Aminotransferase 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for alanine aminotransferase measurement.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
U/L | 1.3 (10.1) | 0.9 (9.0) | 0.6 (11.6)

36. Secondary Outcome: Change From Baseline in Albumin 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for albumin measurement.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
g/dL | -0.02 (0.25) | -0.05 (0.25) | -0.03 (0.25)

37. Secondary Outcome: Change From Baseline in Alkaline Phosphatase 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for alkaline phosphatase measurement.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
U/L | 2.1 (18.9) | 1.4 (12.3) | -0.2 (14.4)

38. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for aspartate aminotransferase measurement.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 339
U/L | -0.0 (9.5) | -0.1 (9.4) | -0.3 (13.3)

39. Secondary Outcome: Change From Baseline in Total Bilirubin 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for total bilirubin measurement.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
umol/L | -0.1 (3.3) | -0.2 (3.9) | -0.2 (3.3)

40. Secondary Outcome: Change From Baseline in Potassium 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for potassium measurement.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 339
mmol/L | 0.01 (0.43) | 0.04 (0.42) | 0.04 (0.43)

41. Secondary Outcome: Change From Baseline in Creatinine 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for creatinine measurement.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
umol/L | 2.0 (8.8) | 1.8 (7.5) | 1.8 (15.6)

42. Secondary Outcome: Change From Baseline in Total Protein 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for total protein measurement.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
g/dL | 0.03 (0.40) | 0.02 (0.37) | -0.02 (0.36)

43. Secondary Outcome: Change From Baseline in Urinary Albumin-to-creatinine Ratio 26 Weeks After Randomisation
Description: as for outcome 30
Time Frame: Week 0, week 26
Population: Analysis was based on the safety analysis set. Number of participants analysed=participants with available data for urinary albumin and creatinine measurement.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 339 | 340
mg/mmol | 0.636 (7.361) | -0.379 (11.095) | 0.656 (12.739)

44. Secondary Outcome: Change From Baseline in Urinalysis (Ketones) 26 Weeks After Randomisation
Description: Presence of ketone in urine was assessed by urine dipstick and categorised as: Negative, Positive, Trace, 1+, 2+, 3+. Change from baseline is represented in terms of percentage of patients with ketone values at week 0 and week 26 (last on-treatment value). Last on-treatment value contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number analysed=number of subjects with available data for ketones values.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Week 0: Negative | 96.2 | 97.1 | 92.7
  Week 0: Positive | 0.0 | 0.0 | 0.0
  Week 0: Trace | 2.0 | 1.8 | 5.3
  Week 0: 1+ | 1.8 | 1.2 | 1.8
  Week 0: 2+ | 0.0 | 0.0 | 0.3
  Week 0: 3+ | 0.0 | 0.0 | 0.0
  Last on-treatment value: Negative: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: Negative | 92.3 | 89.7 | 90.0
  Last on-treatment value:Positive: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value:Positive | 0.0 | 0.0 | 0.0
  Last on-treatment value: Trace: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: Trace | 5.0 | 6.5 | 6.5
  Last on-treatment value:1+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value:1+ | 2.1 | 3.2 | 2.9
  Last on-treatment value: 2+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: 2+ | 0.6 | 0.6 | 0.6
  Last on-treatment value: 3+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: 3+ | 0.0 | 0.0 | 0.0

45. Secondary Outcome: Change From Baseline in Urinalysis (Protein) 26 Weeks After Randomisation
Description: Presence of protein in urine was assessed by urine dipstick and categorised as: Negative, Positive, Trace, 1+, 2+, 3+. Change from baseline is represented in terms of percentage of patients with protein values at week 0 and week 26 (last on-treatment value). Last on-treatment value contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number analysed=number of subjects with available data for protein values.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Week 0: Negative | 82.2 | 79.5 | 80.4
  Week 0: Positive | 0.0 | 0.0 | 0.0
  Week 0: Trace | 12.0 | 14.4 | 13.5
  Week 0: 1+ | 4.4 | 4.1 | 3.5
  Week 0: 2+ | 1.2 | 1.2 | 2.0
  Week 0: 3+ | 0.3 | 0.9 | 0.6
  Last on-treatment value: Negative: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: Negative | 83.5 | 82.6 | 78.8
  Last on-treatment value:Positive: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value:Positive | 0.0 | 0.0 | 0.0
  Last on-treatment value: Trace: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: Trace | 8.6 | 10.9 | 12.4
  Last on-treatment value:1+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value:1+ | 5.9 | 4.7 | 6.5
  Last on-treatment value: 2+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: 2+ | 1.5 | 1.2 | 2.1
  Last on-treatment value: 3+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: 3+ | 0.6 | 0.6 | 0.3

46. Secondary Outcome: Change From Baseline in Urinalysis (Erythrocytes) 26 Weeks After Randomisation
Description: Presence of erythrocytes in urine was assessed by urine dipstick and categorised as: Negative, Positive, Trace, 1+, 2+, 3+. Change from baseline is represented in terms of percentage of patients with erythrocytes values at week 0 and week 26 (last on-treatment value). Last on-treatment value contains the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number analysed=number of subjects with available data for erythrocytes values.
Measure: Number; unit: percentage of subjects
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
percentage of subjects
  Week 0: Negative | 95.3 | 93.3 | 93.3
  Week 0: Positive | 0.0 | 0.0 | 0.0
  Week 0: Trace | 1.8 | 2.3 | 3.2
  Week 0: 1+ | 0.9 | 1.5 | 2.0
  Week 0: 2+ | 1.2 | 0.9 | 0.6
  Week 0: 3+ | 0.9 | 2.1 | 0.9
  Last on-treatment value: Negative: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: Negative | 93.5 | 91.7 | 91.8
  Last on-treatment value:Positive: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value:Positive | 0.0 | 0.0 | 0.0
  Last on-treatment value: Trace: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: Trace | 2.7 | 3.8 | 2.6
  Last on-treatment value:1+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value:1+ | 1.5 | 0.9 | 2.1
  Last on-treatment value: 2+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: 2+ | 0.6 | 2.1 | 1.8
  Last on-treatment value: 3+: number analyzed (Participants) | 339 | 339 | 340
  Last on-treatment value: 3+ | 1.8 | 1.5 | 1.8

47. Secondary Outcome: Change From Baseline in Anti-insulin Aspart (Specific and Cross-reacting With Human Insulin) Antibody Development 26 Weeks After Randomisation
Description: Insulin aspart antibody titres (antibodies specific for insulin aspart and those cross-reacting with human insulin) measured at baseline and at 26 weeks. Week 26 data are based on the last on-treatment value which contains the last available measurement in the on-treatment period. Anti-insulin aspart antibody was measured as % bound radioactivity-labelled insulin aspart/Total added radioactivity-labelled insulin aspart (%B/T).
Time Frame: Week 0, week 26
Population: Analysis was based on the SAS. Number analysed=number of subjects with available data for anti-insulin aspart antibody.
Measure: Mean (Standard Deviation); unit: % B/T
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 342 | 341 | 342
% B/T
  Anti-insulin aspart specific antibodies: number analyzed (Participants) | 337 | 333 | 333
  Anti-insulin aspart specific antibodies | 0.033 (0.777) | -0.027 (1.077) | -0.013 (1.568)
  Cross-reacting to human insulin: number analyzed (Participants) | 337 | 334 | 332
  Cross-reacting to human insulin | -0.972 (6.028) | -1.799 (6.812) | -1.427 (5.527)

48. Secondary Outcome: Change From Baseline in Body Weight 26 Weeks After Randomisation
Description: The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number of subjects analysed=subject with data available for body weight.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
kg | 1.43 (2.66) | 1.14 (2.95) | 1.24 (2.60)

49. Secondary Outcome: Change From Baseline in Body Mass Index 26 Weeks After Randomisation
Description: as for outcome 48
Time Frame: Week 0, week 26
Population: Analysis was based on SAS. Number of subjects analysed=subject with data available for body mass index.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 340 | 340 | 340
kg/m^2 | 0.49 (0.91) | 0.39 (1.02) | 0.43 (0.89)

ADVERSE EVENTS:
Time Frame: Week 0 to week 26 (+7 days)
Description: A TEAE was defined as an event that had an onset date on or after the first day of exposure to randomised treatment, and no later than seven days after the last day of randomised treatment.
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
All-Cause Mortality (participants affected / at risk) | 0/342 | 0/341 | 0/342
Serious Adverse Events (participants affected / at risk) | 20/342 | 17/341 | 17/342
Other Adverse Events (participants affected / at risk) | 154/342 | 152/341 | 161/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (Meal) (N=342) | Faster Aspart (Post) (N=341) | NovoRapid (Meal) (N=342)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Collagen disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (8) | 3 (6) | 6 (6)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (Meal) (N=342) | Faster Aspart (Post) (N=341) | NovoRapid (Meal) (N=342)
Blood glucose decreased (Investigations) | 58 (81) | 67 (83) | 68 (82)
Influenza (Infections and infestations) | 21 (22) | 14 (14) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 30 (38) | 26 (34) | 27 (34)
Viral upper respiratory tract infection (Infections and infestations) | 73 (101) | 70 (100) | 80 (118)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02500706/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02500706/SAP_001.pdf